CLINICAL TRIAL: NCT05350423
Title: Use of Urinary Biomarkers to Quantify Degree of Renal, Parenchymal and Urothelial Damage During Ureteroscopy
Brief Title: Trial Assessing Renal Damage During Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mantu Gupta, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-21-00084; GCO# 21-0054 (Other Grant/Funding Number: New York Academy of Medicine)
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Thulium Fibre Laser (TFL) (Experimental): Patients who are randomized to undergo ureteroscopic laser lithotripsy with the Thulium fibre laser (TFL)
  Interventions: Device: Thulium Fibre Laser
- Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) (Experimental): Patients who are randomized to undergo ureteroscopic laser lithotripsy with the Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) laser
  Interventions: Device: Holmium:Yttrium-Aluminum-Garnet

INTERVENTIONS:
Device: Thulium Fibre Laser — The TFL is a relatively new laser in the field of urology. First introduced on the market in 2017, it offers theoretically superior stone dusting qualities and smaller fiber sizes to allow for better irrigation.
  Other Names: TFL
  Arms: Thulium Fibre Laser (TFL)
Device: Holmium:Yttrium-Aluminum-Garnet — The Ho:YAG is currently the most commonly used laser in the field of urology and for the better part of the last 3 decades has been considered the gold standard for laser lithotripsy.
  Other Names: Ho:YAG
  Arms: Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)

SUMMARY:
This is an ongoing randomized controlled trial of patients undergoing URSLL with unilateral non-obstructing renal stones. Patients are randomized to undergo URSLL with either the TFL or Ho:YAG laser. Each patient's urine is collected immediately pre-op (V1), 1 hour post-op (V2), and 10 days post-op (POD#10, V3). Samples are analyzed by enzyme-linked immunosorbent assay (ELISA) for the following biomarkers: Kidney injury molecule-1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL), and β2-microglobulin (β2M), then normalized to urine creatinine.

DETAILED DESCRIPTION:
Patients scheduled for ureteroscopic laser lithotripsy (URSLL) will be screened and if eligible and agreeable, enrolled into the study. Patients will then be randomized preoperatively via block randomization in groups of 5 to receive lithotripsy with either Ho:YAG or TFL laser intraoperatively. All patients enrolled will have a ureteral stent placed at the end of the procedure.

After induction of anesthesia but before any surgical intervention, the surgeon will empty the bladder and collect a sample of urine that will serve as the "Preoperative Urine Sample". One hour following the end of the procedure, a second sample of urine will be collected from the Foley catheter that will serve as the "Immediate Post-Op Urine Sample". A third and final urine sample of urine will be collected approximately 10 days postoperatively just prior to stent removal and serve as the "Follow-up urine sample". Patients for whom all three urine specimens are collected will be considered to have completed the study. Immediately after collection, the samples will be stored in a freezer at -80 ºC. All samples will be analyzed for biomarkers of renal parenchymal injury to determine differences between pre- and postoperative concentrations. The biomarkers that will be quantified include Kidney Injury Molecule-1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL), and Beta-2-microglobulin (B2M).

Concentrations of urinary biomarkers are determined in duplicate from urine samples using the multiplex cytokine panel [MILLIPLEX MAP Human Kidney Injury Panel 1 (KIM-1), Panel 2 (N-GAL2) and Panel 3 (B2 microglobulin)- Millipore Corp., Burlington, MA] as per manufacturer's instructions. The urine samples were 1:2 diluted for Panel 1, 1:100 diluted for Panel 2 and 1:500 diluted for Panel 3. The kit provided lyophilized pre-mixed standard was reconstituted and used to generate 6-point serial dilutions and run on assay plate along with the samples. Analyte median fluorescent intensity (MFI) values were obtained.

Anticipate enrollment is 108 patients total (54 in each cohort) to adequately power the study based upon an alpha of 0.05 statistical power of 0.80.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patients undergoing unilateral ureteroscopic laser lithotripsy for the treatment of non-obstructing renal stones
* Total stone burden between 5 and 20 mm

Exclusion Criteria:

* Presence of pre-existing indwelling ureteral stent
* Presence of hydronephrosis preoperatively (on either side)
* CKD as defined by eGFR < 60 mL/min
* GU anatomical anomalies (including urinary diversion, solitary kidney, ureteral stricture disease, ureteropelvic junction obstruction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mantu Gupta, Principal Investigator — Department of Urology, Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All data will be presented/shared as aggregates.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Started | 54 | 54
Completed | 46 | 45
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 3 | 3
Not completed — screen failure | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.0 [46.5 to 63.5] | 56.0 [39.0 to 67.5] | 57.5 [42.5 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 23 | 18 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 10 | 26
  Not Hispanic or Latino | 29 | 34 | 63
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 38 | 33 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Kidney Injury Molecule-1 (KIM-1)
Description: Urinary biomarker - a specific biomarker of renal damage to measure the degree of renal parenchymal damage.
Time Frame: Baseline, 1 hour postoperatively, and 10 days postoperatively
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 46 | 45
ng/ml
  Baseline | 0.01077 (0.0087) | 0.01228 (0.0124)
  1 hour post-op | 0.0246 (0.0243) | 0.02413 (0.0229)
  10 days post-op | 0.0161 (0.0127) | 0.0188 (0.0118)

2. Primary Outcome: Change in Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: Urinary biomarker - a specific biomarker of renal damage to measure the degree of renal parenchymal damage.
Time Frame: Baseline, 1 hour postoperatively, and 10 days postoperatively
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 46 | 45
ng/ml
  baseline | 0.5263 (0.9338) | 0.5723 (1.4454)
  1 hour post-op | 2.5181 (4.4884) | 2.4486 (4.6525)
  10 days post-op | 1.8233 (2.4811) | 2.4499 (6.8280)

3. Primary Outcome: Change in β2-microglobulin (β2M)
Description: Urinary biomarker - a specific biomarker of renal damage to measure the degree of renal parenchymal damage.
Time Frame: Baseline, 1 hour postoperatively, and 10 days postoperatively
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 46 | 45
ng/ml
  baseline | 2.1262 (3.5700) | 2.7747 (6.5284)
  1 hour post-op | 25.6231 (96.8722) | 17.1472 (42.5166)
  10 days post-op | 12.5832 (54.7001) | 4.4599 (14.0700)

4. Secondary Outcome: Operative Time
Description: Operative time (minutes) is calculated from time of procedure start (insertion of endoscope into urethral meatus) to time of removal of endoscope from urethral meatus after procedure completion.
Time Frame: Day 1, Intraoperatively
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 46 | 45
minutes | 52.5 [42.8 to 72.3] | 56.0 [42.0 to 68.0]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05350423/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05350423/ICF_001.pdf